CLINICAL TRIAL: NCT04787874
Title: Effect of Health Habits on Outcomes in Plastic and Reconstructive Surgery
Brief Title: Effect of Prehabilitation on Surgical Outcomes of Abdominally-based Plastic Surgery Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cara Black, Resident Physician, PGY-1, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60419
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Ventral Hernia; Panniculus; Abdominoplasty; Flap Reconstruction
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control arm will receive no additional prehabilitation material prior to material. Rather, they will receive standard preoperative care in which they will be given standard advice on nutrition and fitness. REDcap surveys will be administered.
- Prehab Intervention Arm (Experimental): The intervention arm will receive access to the prehab program (abdominal workout videos) and surveys via RedCAP.The program will start no less than 14 days before the date of surgery.
  Interventions: Behavioral: Prehabilitation Program

INTERVENTIONS:
Behavioral: Prehabilitation Program — Nutrition component: Participants will receive information on how to follow a healthy diet (Mediterranean-style diet) with emphasis on whole foods, plants, lean protein, olive oil; restriction of red meats, processed meats, processed foods, added sugar)
  Exercise component: Participants will receive an activity tracker to use during the study period (3+ weeks before surgery, and 30 days after surgery). Participants will be assigned strength exercises to work on core strength and proximal muscle strength (biceps/triceps, quads, hamstrings, calves).The exercises will mainly be focused on strengthening the abdominal wall. Exercises will be tailored to patients' individual capabilities. They will also be assigned cardio exercises - either low-intensity steady state cardio vs High Intensity Interval training. Level of cardio exercise will be tailored based on patient's Duke Activity score and baseline activity.
  Arms: Prehab Intervention Arm

SUMMARY:
The purpose of this study is to determine whether a program to optimize patient physical fitness and nutrition ("prehabilitation") prior to and after plastic surgery involving the abdomen improves surgical outcomes. The investigators hope to determine how a multimodal peri-operative prehabilitation program can be most effective in engaging and motivating patients to physically and mentally get ready for an abdominally-based plastic surgery operation. The overall goal is to determine if this program will improve post-operative recovery after abdominally-based plastic surgery. The importance of this new knowledge is better understanding of ways that plastic surgeons can improve outcomes, engagement, and experience of patients undergoing abdominally-based plastic surgery operations. This would translate to increased healthcare value and better long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients (>18 years) who are undergoing elective abdominally-based plastic surgery operations in 3+ weeks by one of the following plastic surgeons: Nazerali, Lee, Murphy, Nguyen, Lorenz.

Exclusion Criteria:

* Patients who do not speak English
* Patients who do not have access to a smartphone or internet/cell service.
* Patients who are undergoing another intervention study that consists of a nutrition and/or exercise behavior change.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2025-05-23 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of surgical complications (Post-op days 7-14) | Post-operative days 7-14
  Will analyze the occurrence of surgical complications after surgery. Hematoma, seroma, or abscess.
Occurrence of surgical complications (Post-op day 30) | Post-operative day 30
  Will analyze the occurrence of surgical complications after surgery. Hematoma, seroma, or abscess.
Occurrence of surgical complications (Post-op day 90) | Post-operative day 90
  Will analyze the occurrence of surgical complications after surgery. Hematoma, seroma, or abscess.
Occurrence of surgical complications (Post-op day 180) | Post-operative day 180
  Will analyze the occurrence of surgical complications after surgery. Hematoma, seroma, or abscess.
Occurrence of surgical complications (Post-op day 360) | Post-operative day 360
  Will analyze the occurrence of surgical complications after surgery. Hematoma, seroma, or abscess.
Patient-Reported Outcome Measures: RAND 36-Item Health Survey (RAND-36) on Post-op days 7-14 | Post-operative days 7-14
  Will use the RAND 36-Item Health Survey (RAND-36) to assess the patient's perceived health following their surgical procedure. The score for RAND-36 ranges from 0-100, having higher scores mean better outcomes.
Patient-Reported Outcome Measures: Abdominal Surgery Impact Scale (ASIS) on Post-op days 7-14 | Post-operative days 7-14
  Will use the Abdominal Surgery Impact Scale (ASIS) to assess the patient's perceived health following their surgical procedure. The ASIS score ranges from 18-126, having higher scores indicate better quality of life.
Patient-Reported Outcome Measures: RAND 36-Item Health Survey (RAND-36) on Post-op day 30 | Post-operative day 30
  Will use the RAND 36-Item Health Survey (RAND-36) to assess the patient's perceived health following their surgical procedure. The score for RAND-36 ranges from 0-100, having higher scores mean better outcomes.
Patient-Reported Outcome Measures: Abdominal Surgery Impact Scale (ASIS) on Post-op day 30 | Post-operative day 30
  Will use the Abdominal Surgery Impact Scale (ASIS) to assess the patient's perceived health following their surgical procedure. The ASIS score ranges from 18-126, having higher scores indicate better quality of life.
Patient-Reported Outcome Measures: RAND 36-Item Health Survey (RAND-36) on Post-op day 90 | Post-operative day 90
  Will use the RAND 36-Item Health Survey (RAND-36) to assess the patient's perceived health following their surgical procedure. The score for RAND-36 ranges from 0-100, having higher scores mean better outcomes.
Patient-Reported Outcome Measures: Abdominal Surgery Impact Scale (ASIS) on Post-op day 90 | Post-operative day 90
  Will use the Abdominal Surgery Impact Scale (ASIS) to assess the patient's perceived health following their surgical procedure. The ASIS score ranges from 18-126, having higher scores indicate better quality of life.
Patient-Reported Outcome Measures: RAND 36-Item Health Survey (RAND-36) on Post-op day 180 | Post-operative day 180
  Will use the RAND 36-Item Health Survey (RAND-36) to assess the patient's perceived health following their surgical procedure. The score for RAND-36 ranges from 0-100, having higher scores mean better outcomes.
Patient-Reported Outcome Measures: Abdominal Surgery Impact Scale (ASIS) on Post-op day 180 | Post-operative day 180
  Will use the Abdominal Surgery Impact Scale (ASIS) to assess the patient's perceived health following their surgical procedure. The ASIS score ranges from 18-126, having higher scores indicate better quality of life.
Patient-Reported Outcome Measures: RAND 36-Item Health Survey (RAND-36) on Post-op day 360 | Post-operative day 360
  Will use the RAND 36-Item Health Survey (RAND-36) to assess the patient's perceived health following their surgical procedure. The score for RAND-36 ranges from 0-100, having higher scores mean better outcomes.
Patient-Reported Outcome Measures: Abdominal Surgery Impact Scale (ASIS) on Post-op day 360 | Post-operative day 360
  Will use the Abdominal Surgery Impact Scale (ASIS) to assess the patient's perceived health following their surgical procedure. The ASIS score ranges from 18-126, having higher scores indicate better quality of life.
Physical Function Test: 6-minute walk test at Time of Enrollment | Time of enrollment
  Will use the 6-minute walk test. The 6-minute walk test will be used to assess aerobic capacity and endurance. A normal walk distance ranges from 400 to 700 m.
Physical Function Test: 5-times-sit-to-stand test at Time of Enrollment | Time of enrollment
  Will use the 5-times-sit-to-stand test. The 5-times-sit-to-stand test is a method to quantify functional lower extremity strength. Lower times indicate better scores.
Physical Function Test: Timed-up-and-go test at Time of Enrollment | Time of enrollment
  Will use the timed-up-and-go test. The timed-up-and go test assesses one's mobility. A lower score signifies better mobility.
Physical Function Test: 6-minute walk test at 3 weeks | 3 weeks
  Will use the 6-minute walk test. The 6-minute walk test will be used to assess aerobic capacity and endurance. A normal walk distance ranges from 400 to 700 m.
Physical Function Test: 5-times-sit-to-stand test at 3 weeks | 3 weeks
  Will use the 5-times-sit-to-stand test. The 5-times-sit-to-stand test is a method to quantify functional lower extremity strength. Lower times indicate better scores.
Physical Function Test: Timed-up-and-go test at 3 weeks | 3 weeks
  Will use the timed-up-and-go test. The timed-up-and go test assesses one's mobility. A lower score signifies better mobility.
Physical Function Test: 6-minute walk test on Post-op Day 30 | Post-operative day 30
  Will use the 6-minute walk test. The 6-minute walk test will be used to assess aerobic capacity and endurance. A normal walk distance ranges from 400 to 700 m.
Physical Function Test: 5-times-sit-to-stand-test on Post-op Day 30 | Post-operative day 30
  Will use the 5-times-sit-to-stand test. The 5-times-sit-to-stand test is a method to quantify functional lower extremity strength. Lower times indicate better scores.
Physical Function Test: Timed-up-and-go test on Post-op Day 30 | Post-operative day 30
  Will use the timed-up-and-go test. The timed-up-and go test assesses one's mobility. A lower score signifies better mobility.
Physical Function Test: 6-minute walk test on Post-op Day 90 | Post-operative day 90
  Will use the 6-minute walk test. The 6-minute walk test will be used to assess aerobic capacity and endurance. A normal walk distance ranges from 400 to 700 m.
Physical Function Test: 5-times-sit-to-stand test on Post-op Day 90 | Post-operative day 90
  Will use the 5-times-sit-to-stand test. The 5-times-sit-to-stand test is a method to quantify functional lower extremity strength. Lower times indicate better scores.
Physical Function Test: Timed-up-and-go test on Post-op Day 90 | Post-operative day 90
  Will use the timed-up-and-go test. The timed-up-and go test assesses one's mobility. A lower score signifies better mobility.

SECONDARY OUTCOMES:
Change from Baseline Albumin Levels at Time of Surgery | Enrollment to time of surgery
  To analyze nutritional status
Change from Baseline Prealbumin Levels at Time of Surgery | Enrollment to time of surgery
  To analyze nutritional status
Change from Baseline Transferrin Levels at Time of Surgery | Enrollment to time of surgery
  To analyze nutritional status
Change from Baseline C-reactive Protein Levels at Time of Surgery | Enrollment to time of surgery
  To analyze level of physiologic inflammation
Change from Baseline Erythrocyte Sedimentation Rates at Time of Surgery | Enrollment to time of surgery
  To analyze level of physiologic inflammation
Change from Baseline Hemoglobin A1C Levels at Time of Surgery | Enrollment to time of surgery
  To analyze degree of diabetes mellitus control
Change from Baseline Plasma Glucose Levels at Time of Surgery | Enrollment to time of surgery
  To analyze degree of diabetes mellitus control
Change from Baseline White Blood Cell Count at Time of Surgery | Enrollment to time of surgery
  Assessment for leukocytosis, anemia, renal disease; Part of the complete blood count.
Change from Baseline Hemoglobin Levels at Time of Surgery | Enrollment to time of surgery
  Assessment for leukocytosis, anemia, renal disease; Part of the complete blood count.
Change from Baseline Hematocrit Levels at Time of Surgery | Enrollment to time of surgery
  Assessment for leukocytosis, anemia, renal disease; Part of the complete blood count.
Change from Baseline Platelet Levels at Time of Surgery | Enrollment to time of surgery
  Assessment for leukocytosis, anemia, renal disease; Part of the complete blood count.
Change from Baseline Chloride Levels at Time of Surgery | Enrollment to time of surgery
  Assessment for leukocytosis, anemia, renal disease; Part of Basic Metabolic Panel
Change from Baseline Sodium Levels at Time of Surgery | Enrollment to time of surgery
  Assessment for leukocytosis, anemia, renal disease; Part of Basic Metabolic Panel
Change from Baseline Potassium Levels at Time of Surgery | Enrollment to time of surgery
  Assessment for leukocytosis, anemia, renal disease; Part of Basic Metabolic Panel
Change from Baseline Carbon Dioxide Levels at Time of Surgery | Enrollment to time of surgery
  Assessment for leukocytosis, anemia, renal disease; Part of Basic Metabolic Panel
Change from Baseline Blood Urea Nitrogen Levels at Time of Surgery | Enrollment to time of surgery
  Assessment for leukocytosis, anemia, renal disease; Part of Basic Metabolic Panel
Change from Baseline Creatinine Levels at Time of Surgery | Enrollment to time of surgery
  Assessment for leukocytosis, anemia, renal disease; Part of Basic Metabolic Panel
Change from Baseline Blood Glucose Levels at Time of Surgery | Enrollment to time of surgery
  Assessment for leukocytosis, anemia, renal disease; Part of Basic Metabolic Panel

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Kin, MD, Study Director — Asst Prof-Med Ctr Line; Cara Black, MD, Principal Investigator — Resident
Locations (2):
- United States (2):
  - Stanford Cancer Center South Bay, San Jose, California
  - Stanford Plastic and Reconstructive Surgery Clinic, Stanford, California

IPD SHARING:
Plan to Share IPD: No